CLINICAL TRIAL: NCT00003573
Title: A Phase I/II Feasibility Study of Oral Etoposide Given Concurrently With Radiotherapy Followed With Dose Intensive Adjuvant Chemotherapy for Children With Newly Diagnosed High Stage Medulloblastoma
Brief Title: Etoposide Plus Radiation Therapy Followed by Combination Chemotherapy in Treating Children With Newly Diagnosed Advanced Medulloblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9631; POG-9631 (Other: Pediatric Oncology Group); CDR0000066640 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Brain Tumors; Central Nervous System Tumors
Keywords: untreated childhood medulloblastoma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cisplatin; Cyclophosphamide; Etoposide; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment 1, Etoposide, 50mg/m2/day (Experimental): Patients begin treatment within 1 month of surgery. Patients receive 6 weeks of radiation therapy to the head and spine, with boosts to the posterior fossa and to sites of metastasis. Patients also receive 2 courses of oral etoposide once daily for 3 weeks concurrent with and immediately following radiotherapy (weeks 1-3 and 5-7).
  Patients then receive adjuvant chemotherapy consisting of cisplatin IV once every 4 weeks for 3 courses beginning on week 11, oral etoposide daily for 21 days every 4 weeks for 3 courses (weeks 11, 15, and 19), cyclophosphamide IV on days 1 and 2 with filgrastim (G-CSF) SQ daily for at least 10 days every 4 weeks for 8 courses (weeks 23-51), and vincristine IV on days 1, 8, and 15 every 4 weeks for 8 courses (weeks 23-51).
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: cyclophosphamide; Drug: etoposide; Drug: vincristine sulfate; Radiation: radiation therapy
- Treatment 2, Etoposide, 35mg/m2/day (Experimental): Patients begin treatment within 1 month of surgery. Patients receive 6 weeks of radiation therapy to the head and spine, with boosts to the posterior fossa and to sites of metastasis. Patients also receive 2 courses of oral etoposide once daily for 3 weeks concurrent with and immediately following radiotherapy (weeks 1-3 and 5-7).
  Patients then receive adjuvant chemotherapy consisting of cisplatin IV once every 4 weeks for 3 courses beginning on week 11, oral etoposide daily for 21 days every 4 weeks for 3 courses (weeks 11, 15, and 19), cyclophosphamide IV on days 1 and 2 with filgrastim (G-CSF) SQ daily for at least 10 days every 4 weeks for 8 courses (weeks 23-51), and vincristine IV on days 1, 8, and 15 every 4 weeks for 8 courses (weeks 23-51).
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: cyclophosphamide; Drug: etoposide; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen®; NSC #614629
Drug: cisplatin
  Other Names: Cis-diamminedichloroplatinum II; CDDP; Platinol; NSC #119875
Drug: cyclophosphamide
  Other Names: CTX; Cytoxan; NSC #026271; IND #7089
Drug: etoposide
  Other Names: VP-16; VePesid; NSC #141540; IND #9197
Drug: vincristine sulfate
  Other Names: VCR; Oncovin; NSC #067574; IND #7161
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of etoposide plus radiation therapy followed by combination chemotherapy in treating children with newly diagnosed advanced medulloblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the response rate and toxicity of oral etoposide and radiotherapy in children with newly diagnosed high stage medulloblastoma.
* Compare the response rate and toxicity of these patients to historical control patients registered on POG #9031.
* Estimate the 2-year event-free survival and overall survival of these patients.
* Evaluate the toxicity of dose intensive chemotherapy with oral etoposide, cisplatin, cyclophosphamide, and vincristine following craniospinal irradiation in these patients.

OUTLINE: Patients begin treatment within 1 month of surgery. Patients receive 6 weeks of radiotherapy to the head and spine, with boosts to the posterior fossa and to sites of metastasis. Patients also receive 2 courses of oral etoposide once daily for 3 weeks concurrent with and immediately following radiotherapy (weeks 1-3 and 5-7).

Patients then receive adjuvant chemotherapy consisting of cisplatin IV once every 4 weeks for 3 courses beginning on week 11, oral etoposide daily for 21 days every 4 weeks for 3 courses (weeks 11, 15, and 19), cyclophosphamide IV on days 1 and 2 with filgrastim (G-CSF) SQ daily for at least 10 days every 4 weeks for 8 courses (weeks 23-51), and vincristine IV on days 1, 8, and 15 every 4 weeks for 8 courses (weeks 23-51).

Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and annually thereafter.

PROJECTED ACCRUAL: A total of 48 patients will be accrued for this study within about 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically diagnosed advanced (high grade) childhood medulloblastoma
* Residual disease of at least 1.5 cm2 in size on MRI or CT scan OR
* Evidence of CNS or extraneural metastases

PATIENT CHARACTERISTICS:

Age:

* 3 to 21

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* SGPT less than 5 times normal
* Bilirubin less than 1.5 mg/dL

Renal:

* Creatinine less than 1.7 mg/dL OR
* Creatinine clearance greater than 70 mL/min

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior corticosteroids allowed

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 1998-11; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of oral etoposide at 50 mg/m2/day given concurrently with radiotherapy followed with dose intensive adjuvant chemotherapy in children with newly diagnosed high stage medulloblastoma | End of course 1 (week 10)
  It is possible that unacceptably high levels of toxicity may arise. For this reason, there is a 3-stage stopping rule designed to allow the Study Coordinator to stop this study early if it appears that the true proportion of eligible patients who suffer unacceptable levels of toxicity exceeds 10%.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Moghrabi, MD, Study Chair — Hopital Sainte Justine
Locations (106):
- United States (94):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Children's Hospital and Health Center, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - CCOP - Florida Pediatric, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Portland, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. John's Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - James H. Quillen College of Medicine, Johnson City, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - MBCCOP - South Texas Pediatric, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Clinic, Temple, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Carilion Roanoke Community Hospital, Roanoke, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Medical School-Charleston, Charleston, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- San Jorge Childrens Hospital, Santurce, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Clinique de Pediatrie, Geneva

REFERENCES:
- [Derived] Tarbell NJ, Friedman H, Polkinghorn WR, Yock T, Zhou T, Chen Z, Burger P, Barnes P, Kun L. High-risk medulloblastoma: a pediatric oncology group randomized trial of chemotherapy before or after radiation therapy (POG 9031). J Clin Oncol. 2013 Aug 10;31(23):2936-41. doi: 10.1200/JCO.2012.43.9984. Epub 2013 Jul 15. PMID 23857975